CLINICAL TRIAL: NCT03495310
Title: Effect of Mindfulness on Some Hormones That Regulate Stress and Appetite, and on the Body Weight of Obese Schoolchildren. Controlled Clinical Trial
Brief Title: Effect of Mindfulness on Stress, Appetite Hormones and Body Weight of Obese Schoolchildren. Controlled Clinical Trial
Acronym: Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Mardia Guadalupe Lopez Alarcon, Dr. Mardia Lopez-Alarcon, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2017-785-096
Record Dates: First submitted 2018-03-06; First posted 2018-04-12 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Obesity, Childhood; Mindfulness
MeSH Terms: conditions — Pediatric Obesity | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): In this group, children and their parents will receive a mindfulness session once a week, with a duration of 90 minutes, during 8 weeks (sessions will be separated for children and parents). Mindfulness sessions will be coordinated by experts in mindfulness techniques in children and adults respectively from the collaborator Institution "Spanish School of Transpersonal Development" Previous to the session, a 24-hour food recall questionnaire will be applied to offer a meal plan restricted in 500 kcal. The 24-R will be repeated at each session in order to make adjustments to the meal plan if necessary. Also a 60-minute walk 3 times a week will be recommended
  Interventions: Behavioral: Mindfulness
- Control (No Intervention): In this group, children and their parents will receive information regarding what is a healthy diet and physical activity attached to the World Health Organization recommendations. The session will be coordinated by a pediatric endocrinologist. Previous to the session, a 24-hour food recall questionnaire will be applied to offer a meal plan restricted in 500 kcal. The 24-R will be repeated at each session in order to make adjustments to the meal plan when necessary. Also a 60-minute walk 3 times a week will be recommended

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness is a method based on the concentration of attention, awareness and meditation, which has been used successfully to reduce stress, depression and anxiety in individuals with some pathology in the short term
  Other Names: method on the concentration of attention
  Arms: Mindfulness

SUMMARY:
In addition to diet and sedentary lifestyle, factors such as stress, depression and anxiety have been found associated in up to 86% of cases of obesity in children. Mindfulness is a method based on the concentration of attention, awareness and meditation, which has been successfully used to reduce stress, depression and anxiety in individuals with some pathology in the short term (eight weeks).

Objective: To determine if an intervention with mindfulness is effective to reduce the stress, appetite, and body weight of a group of school children with obesity and stress comparing them with a group that receives conventional therapy.

Methods For a controlled clinical trial, 60 children of 10-14 years of age with obesity (BMI> 2 SD) and stress (Spence scale> 60) will be selected, and randomly assigned to a group that receives the intervention with mindfulness (M8S), or to the control group (TC);The intervention with Mindfulness will be done once a week for 8 weeks. Measurements of BMI, glucose, leptin, ghrelin, cortisol and insulin will be carried out at the beginning of the study, and repeated at the end of the intervention and eight weeks after finishing the intervention to evaluate relapses.

DETAILED DESCRIPTION:
Parents of children 10-14 years of age with suspected obesity will be invited to participate. When the child and at least one of the parents wish to participate, anthropometry will be performed to calculate the BMI z-score and the Spence questionnaire will be applied to identify stress. If they meet the selection criteria, they will be recorded in a pre-registration form to call them once the sample size is completed in order to start the interventions simultaneously for all the children and in parallel for the two groups.

To initiate the intervention, the children will be summoned in the Research Unit accompanied by at least one of the parents at 7:00 with at least eight hours of fasting, without brushing their teeth and without having performed any physical activity, for explain what their participation in the study consists of and ask them to sign the letters of consent and informed consent. Anthropometric measurements (weight, height, waist circumference) will be taken, and a peripheral blood sample will be taken to determine the concentrations of insulin, glucose, leptin and ghrelin, and a 24-h reminder questionnaire will be applied. When they leave, they will be given a kit for collecting saliva samples to calculate the Cortisol Awakening Response and will be given the appropriate instructions.

Once all the children's anthropometric and diet information has been obtained, they will be randomly assigned to one of the two groups using a computerized random number table. The children assigned to the mindfulness group will be summoned every Wednesday in the classroom of the Research Unit to receive the sessions, which will be taught by an expert in mindfulness techniques in children of the Spanish School of Transpersonal Development. Children assigned to the conventional treatment group will be summoned every Thursday at the same place to receive reinforcement talks aimed at motivating the child and their parents to adhere to the indications of diet and physical activity, taught by a pediatric endocrinologist with nutrition training. involved in the investigation.

Body weight will be measured every week before the session, and biochemical measurements will be repeated at the end of the eight weeks of intervention and eight weeks after the end of the intervention to assess relapses.

ELIGIBILITY:
Inclusion Criteria:

obesity (BMI> 2 SD) and stress (Spence scale> 60) -

Exclusion Criteria:

* taking any antihyperglycemic medication
* obesity of endocrinological origin
* do not wish to participate

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
stress | 8 weeks
  Change in salivary cortisol from baseline to end of intervention

SECONDARY OUTCOMES:
insulin resistance | 8 weeks
  Change in homeostasis model assessment from baseline to the end of intervention
appetite hormones | 8 weeks
  Change in serum ghrelin and leptin from baseline to the end of intervention
weight | 8 weeks
  Change in BMI from baseline to the end of intervention
BMI relapse | 8 weeks
  Change in BMI from the end of intervention to 8 weeks later

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Mardia Lopez Alarcon, Cuauhtémoc, Mexico City
  - Unit or research in Medical Nutrition, Pediatric Hospital CMN "Siglo XXI", Instituto Mexicano del Seguro Social, Mexico City

IPD SHARING:
Plan to Share IPD: No